CLINICAL TRIAL: NCT07022288
Title: A Clinical Study Evaluating the Application of La Roche-Posay's New B5 Multi-Effect Soothing and Repairing Cream on Individuals With Facial Atopic Dermatitis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C25005013
Record Dates: First submitted 2025-05-21; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis of Face

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LA ROCHE-POSAY CICAPLAST BALM (Experimental): Products Application and Usage Instruction
  Mode of application: 0 Day~8 weeks
  Frequency:
  the study participants should apply LA ROCHE-POSAY CICAPLAST BALM to the entire face twice daily (morning and evening), with each application ranging from 0.5 to 0.75 grams.
  Interventions: Other: LA ROCHE-POSAY CICAPLAST BALM, Standard cream
- standard cream (Active Comparator): Products Application and Usage Instruction
  Mode of application: 0 Day~8 weeks
  Frequency:
  the study participants should apply standard cream to the entire face twice daily (morning and evening), with each application ranging from 0.5 to 0.75 grams.
  Interventions: Other: LA ROCHE-POSAY CICAPLAST BALM, Standard cream

INTERVENTIONS:
Other: LA ROCHE-POSAY CICAPLAST BALM, Standard cream — After enrollment, the investigator will generate random serial numbers for grouping through simple randomization.
  LA ROCHE-POSAY CICAPLAST BALM：8 weeks application It is a leave-on product. It should be applied to the face twice a day during the research period.
  Standard cream:8 weeks application It is a leave-on product. It should be applied to the face twice a day during the research period.

SUMMARY:
This study plans to recruit 76 subjects in accordance with the above inclusion and exclusion criteria, with at least 60 subjects completing the study. The study period is 8 weeks, and the subjects need to visit the research center 4 times. After the subjects are enrolled, they will be randomly divided into two groups, including the experimental product group and the control product group.

The physiological indicators of the skin were measured by objective instruments and compared with those of ordinary moisturizers without skin microecological regulation components to evaluate the repair promotion effect and improvement of La Roche-Posay's new B5 Multi-Effect Soothing and Repairing Cream on the affected areas of patients with mild atopic dermatitis on the

ELIGIBILITY:
Inclusion Criteria:

* 1) Chinese males and females aged 18 to 65 years old (including 18 and 65 years old); 2) In good health, without any other chronic diseases or diseases under treatment; 3) Have received atopic dermatitis drug treatments, including but not limited to:

  1. Topical glucocorticoids (TSC), such as 0.05% fluticasone propionate cream, 0.1% mometasone furoate cream, 0.1% hydrocortisone butyrate cream, 0.1% triamcinolone acetonide cream, 0.25% hydrocortisone cream, 0.05% desonide cream/ointment, etc.;
  2. Topical calcineurin inhibitors (TCI), such as 1% pimecrolimus cream, 0.03%/0.1% tacrolimus ointment, etc.;
  3. Oral antihistamines, such as cetirizine hydrochloride tablets, loratadine tablets, ebastine tablets, azelastine hydrochloride tablets, etc.;
  4. Other topical medications, such as zinc oxide oil (paste), black bean distillate oil ointment, topical phosphodiesterase 4 (PDE-4) inhibitor ointment, physiological sodium chloride solution, and other wet dressing medications, etc.; 4) At the baseline visit (Baseline), as determined by a dermatologist:

     * Meeting Yao's diagnostic criteria,
     * Atopic dermatitis severity is mild (Investigator Global Assessment, IGA ≤ 2 points);
     * The condition is in a stable phase and no longer requires topical drug treatment 5) At the baseline visit (Baseline), trans-epidermal water loss (TEWL) measurement value > 15g/m²/h 6) Voluntarily participate in the trial, understand and be willing to sign the informed consent form; 7) Willing to follow the study protocol to use the products provided by the study throughout the study period, not use other similar products, keep diaries, and attend regular follow-ups and other trial requirements.

Exclusion Criteria:

* 1) Study participants who plan to become pregnant, are pregnant, are breastfeeding, are within 6 months after childbirth, or are unwilling to take necessary precautions to avoid pregnancy; 2) Study participants with atopic dermatitis in an acute exacerbation phase; 3) Study participants currently participating in other clinical trials or who have participated in other clinical trials within the past 3 months; 4) Study participants who used functional moisturizers containing skin microecology-regulating ingredients within 1 week before enrollment; 5) Study participants who received physical, chemical, or cosmetic surgical treatments within 3 months before enrollment; 6) Study participants with systemic diseases (severe organ damage), malignant tumors, poorly controlled chronic diseases, acute infectious diseases, major surgeries or trauma, psychological or mental disorders, or who require local or systemic use of drugs/treatments affecting atopic dermatitis due to other diseases; 7) Study participants who experience explosive exacerbation of atopic dermatitis lesions after using the treatment regimen; 8) Study participants with other skin diseases (acne, rosacea, eczema, infections, tumors, etc.) at the study site or other skin conditions interfering with evaluation (birthmarks, scars, etc.); 9) Study participants with a habit of scratching or squeezing atopic dermatitis lesions; 10) Study participants with a history of allergy to the products and related ingredients provided in the study; 11) Study participants with poor compliance, known inability to attend visits on time, or unwillingness to follow the study protocol during the study period; 12) Other circumstances where the investigator deems it inappropriate for the participant to join the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Sebum secretion on the skin surface | Baseline, Time point at 2Week, Time point at 4Week, Time point at 8Week.
  Sebum secretion on the skin surface will be measured by Sebumeter® SM 815 by trained technician.
TEWL on the skin surface | Baseline, Time point immediate,Time point at 2Week, Time point at 4Week, Time point at 8Week.
  TEWL on the skin surface will be measured by Vapometer by trained technician.
Skin hydration on the skin surface | Baseline, Time point immediate,Time point at 2Week, Time point at 4Week, Time point at 8Week.
  Skin hydration on the skin surface will be measured by Corneometer® CM 825 by trained technician.
The pH value of the skin surface | Baseline, Time point immediate,Time point at 2Week, Time point at 4Week, Time point at 8Week.
  The pH value of the skin surface will be measured by Skin-pH Meter PH 905 by trained technician.
Standardized facial image acquisition by VISIA | Baseline,Time point at 2Week, Time point at 4Week, Time point at 8Week.
  Trained professionals will use the standard light source and polarized light source in Visia 7 to photograph the frontal, left, and right sides of the study participants' faces for facial image acquisition.
The safety and tolerability judgment by dermatologists based on the assessment of interviewed symptoms and observed signs | Baseline,Time point at 2Week, Time point at 4Week, Time point at 8Week.
  During the study, dermatologists will assess the facial condition of study participants. At each visit, each participant will be asked: "Are you experiencing any discomfort now?" If the participant answers "yes", the specific type of discomfort (e.g., tightness, stinging, burning, itching, or any other discomfort) should be recorded, along with the intensity and location of the discomfort. Additionally, dermatologists must carefully document the exact location (e.g., left cheek, right cheek, periocular area, etc.) of observed signs (such as erythema, edema, dryness, desquamation, acne, or any other symptoms) during the examination.

SECONDARY OUTCOMES:
The diagnostic criteria for atopic dermatitis evaluated according to Yao's diagnostic criteria | Baseline, Time point immediate,Time point at 2Week, Time point at 4Week, Time point at 8Week.
  Yao's diagnostic evaluation criteria scoring standards are as follows:
  1. Itching;
  2. Typical morphology and location (flexural dermatitis), or atypical morphology and location accompanied by dry skin;
  3. Chronic or chronic relapsing course.
  The diagnosis of atopic dermatitis can be made if all three of the above criteria are met.
The IGA (Investigator Global Assessment) scoring conducted by the investigator | Baseline,Time point at 2Week, Time point at 4Week, Time point at 8Week
  The investigator performs the IGA (Investigator Global Assessment) scoring on the facial condition of study participants.(0 = clear,5 = very severe)
The facial Eczema Area and Severity Index (F-EASI) scoring conducted by the investigator | Baseline,Time point at 2Week, Time point at 4Week, Time point at 8Week
  The Facial Eczema Area and Severity Index (F-EASI) scores erythema (E), edema/induration/papulation (I), excoriation (EX), and lichenification (L) across the entire face, combined with the affected area.
The clinical scoring for facial erythema | Baseline,Time point at 2Week, Time point at 4Week, Time point at 8Week
  The clinical scoring for facial erythema (Erythema) is evaluated by dermatologists using a 0-4 grading scale（0 = none, 4 = severe）.
Study participants perform visual analog scale (VAS) scoring | Baseline, Time point immediate,Time point at 2Week, Time point at 4Week, Time point at 8Week.
  Study participants perform visual analog scale (VAS) scoring for facial Itch, skin tightness, burning, stinging, and pain.
  The Visual Analog Scale (VAS) is a straight line with extreme values of facial discomfort at both ends. The leftmost end of the scale is "no discomfort" (score = 0 mm), and the rightmost end is "extreme discomfort" (the most severe degree imaginable) (score = 100 mm).
The Dermatology Life Quality Index (DLQI) questionnaire completed by study participants | Baseline, Time point at 2Week, Time point at 4Week, Time point at 8Week.
  Study participants fill in the Dermatology Life Quality Index (DLQI) questionnaire based on their actual quality of life.Use a 0-3 scoring scale (0 = none, 3 = very severe).
Skin microbiota detection | Baseline, Time point at 4Week , Time point at 8Week
  Trained operators will sample the marked typical affected areas of atopic dermatitis in study participants for biological sample collection. Microbial samples will be collected using swabs.
  Alpha/beta diversity：Based on next-generation sequencing (NGS) technology, 16S rRNA sequencing will be used to detect changes in skin bacterial species of interest from baseline to time point at 8week, including variations in species richness and diversity (alpha/beta diversity).

CONTACTS AND LOCATIONS:
Overall Officials: Ping Xu, Master, Principal Investigator — Shanghai China-norm Quality Technical Service Co., Ltd.
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No